CLINICAL TRIAL: NCT04217629
Title: Phase I Clinical Study to Evaluate Safety, Tolerance and Pharmacokinetics of SY-005 After Single-dose/Multiple-doses Incremental Intravenous Injection in Healthy Subjects
Brief Title: Single-dose/Multiple-doses Incremental Intravenous Injection of SY-005 （Recombinant Human Annexin A5）in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Yabao Pharmaceutical R&D Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SY005001
Record Dates: First submitted 2020-01-01; First posted 2020-01-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- SY-005 single-dose 0.75mg (Experimental): 4 subjects will be envolved in this group and be injected with 0.75mg of SY-005.
  Interventions: Drug: SY-005
- SY-005 single-dose 2.5mg (Placebo Comparator): This group will be intiated in healthy subjects at a 2.5mg dose. 12 subjects will be envolved in this group and the proportion of subjects injected SY-005 to placebo is 5:1.
  Interventions: Drug: SY-005
- SY-005 single-dose 5mg (Placebo Comparator): This group will be intiated in healthy subjects at a 5mg dose. 12 subjects will be envolved in this group and the proportion of subjects injected SY-005 to placebo is 5:1.
  Interventions: Drug: SY-005
- SY-005 single-dose 10mg (Placebo Comparator): This group will be intiated in healthy subjects at a 10mg dose. 12 subjects will be envolved in this group and the proportion of subjects injected SY-005 to placebo is 5:1.
  Interventions: Drug: SY-005
- SY-005 single-dose 15mg (Placebo Comparator): This group will be intiated in healthy subjects at a 15mg dose. 12 subjects will be envolved in this group and the proportion of subjects injected SY-005 to placebo is 5:1.
  Interventions: Drug: SY-005
- SY-005 single-dose 20mg (Placebo Comparator): This group will be intiated in healthy subjects at a 20mg dose. 12 subjects will be envolved in this group and the proportion of subjects injected SY-005 to placebo is 5:1.
  Interventions: Drug: SY-005
- SY-005 multiple-doses 5mg (Placebo Comparator): This group will be intiated in healthy subjects at a 5mg dose. 10 subjects will be envolved in this group and the proportion of subjects injected SY-005 to placebo is 4:1. The subjects will be injected with SY-005 or placebo for 7days.
  Interventions: Drug: SY-005
- SY-005 multiple-doses 10mg (Placebo Comparator): This group will be intiated in healthy subjects at a 10mg dose. 10 subjects will be envolved in this group and the proportion of subjects injected SY-005 to placebo is 4:1. The subjects will be injected with SY-005 or placebo for 7days.
  Interventions: Drug: SY-005
- SY-005 multiple-doses 20mg (Placebo Comparator): This group will be intiated in healthy subjects at a 20mg dose. 10 subjects will be envolved in this group and the proportion of subjects injected SY-005 to placebo is 4:1. The subjects will be injected with SY-005 or placebo for 7days.
  Interventions: Drug: SY-005

INTERVENTIONS:
Drug: SY-005 — This single-dose group will be initiated in healthy subjects at a 0.75mg dose that is the maximum recommended starting dose(MRSD). Doses will be escalated in subsequent dosing process, after appropriate review of safety data. The subsequent planned doses are2.5mg, 5mg, 10mg, 15mg, 20mg successively. The dose of multiple-doses groups are depending on the results of single-dose groups.

SUMMARY:
This is a single-dose/multiple-doses incremental, randomized, double-blind, parallel, placebo-controlled study on safety, tolerance and pharmacokinetics healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dosed tolerability, pharmacokinetic study of a single-dose/multiple-doses incremental intravenous injection of SY-005（recombinant human annexin A5） in healthy subjects. Six sigle-dose group trials are planned: 0.75mg, 2.5mg, 5mg, 10mg, 15mg,and 20mg and three multiple-doses groups are planned: 5mg, 10mg and 20mg. Single-dose groups are planned to enroll 64 subjects and multiple-doses groups are planned to enroll 30 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-65 (including two values);
* During the screening period, the body weight of male subjects is greater than or equal to 50kg, and that of female subjects is greater than or equal to 45kg, with a body mass index (BMI = weight/height squared (kg/m2)) in the range of 18 to 26 (including both ends);
* Medical history, physical examination, other laboratory examination items and examination related to the test before the test. All the tests were normal or not clinically significant mild abnormalities, clinical research doctors judged that qualified;
* APTT and PT laboratory test results in coagulation function are within the normal range;
* Platelet laboratory examination results are not lower than the lower limit of normal range；
* The venous channel is normal and blood samples can be fully collected according to the plan;
* Subjects must give informed consent to this study before the study and voluntarily sign a written informed consent;
* Subjects are willing to take effective contraceptive measures, and have pregnancy plane during and within 3 months after the stud. Female subjects should be non-lactating, have negative pregnancy test, or have no fertility potential. Women who have been without a uterus for at least 12 months or are considered to have no potential pregnancy.

Exclusion Criteria:

* The subjects are suffering from cardiovascular diseases, respiratory diseases, gastrointestinal diseases, liver and kidney function damage, endocrine diseases, blood system diseases, nervous system diseases, which can significantly change the distribution, metabolism and excretion of test drugs, or the use of test drugs will increase the risk of subjects or affect the analysis of research results;
* QTc interval is not in normal range, male higher than 450 msec and female higher than 470 msec;
* Those who have a history of drug or other allergies, or may be allergic to the study drug or any component of the study drug in the judgment of the researcher;
* Those who completed or withdrawed from a clinical study within 3 months of the screening period, or is currently conducting a clinical study. Or participated in other medical research activities, which the researchers judged unsuitable for this study;
* Have a history of alcohol abuse and drug abuse;
* Those who have donated blood within 3 months, or those who plan to donate blood within 3 months, or those who have transfused blood within 4 weeks before the study;
* Women who consume more than 14 g of alcohol a week and men who consume more than 21 g of alcohol (1 g of alcohol is equivalent to360 mL of beer, 150 mL of wine or 45 mL of liquor) a week;Participants were reluctant to stop drinking between 24 hours before the study began and the end of the study;
* Those who smoke more than 5 cigarettes a day or are unwilling/unable to stop nicotine intake during the study period;
* Abnormal chest X-ray examination with clinical significance;
* 12-lead ecg showed clinically significant abnormalities, and the researcher believed that participating in the experiment would increase the risk of subjects;
* Viral serological evidence during screening: patients with positive hepatitis B surface antigen (HBsAg), positive anti-hcv, or positive anti-HIV antibodyof human immunodeficiency virus (HIV), or positive anti-tp antibody of treponema pallidum;
* Patients who have undergone major surgery within 6 months before drug administration;
* Those who have been screened for the first 4 weeks or plan to receive live vaccines during the trial;
* Fertile eligible subjects (male and female) will not agree to use a reliable contraceptive method (hormone or barrier method or abstinence) during the study period and at least 1 months after administration;
* The sponsor or the investigator decides that the investigator is not suitable to participate in the study; Women who have been without a uterus for at least 12 months or are considered to have no potential pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events of SY-005 | Single-dose: 21 days/ Multiple-doses: 28 days
  Incidence of adverse events of SY-005, collecting number of subjects with adverse events as assessed by CTCAE V5.0. Number of subjects with adverse events, major adverse events, serious adverse events, pregnancy events, abnormal laboratory values, abnormal vital signs, abnormal physical examination, abnormal ECG data.

SECONDARY OUTCOMES:
Area under curve (AUC) of SY-005 following injection of single dose/multiple-doses | Single-dose: 24 hours/ Multiple-doses: 8 days
  To mearsure the study drug concentration in blood samples which collected after injection
Cmax of SY-005 following injection of single dose/multiple-doses | Single-dose: 24 hours/ Multiple-doses: 8 days
  To mearsure the study drug concentration in blood samples which collected after injection
Tmax of SY-005 following injection of single dose | Single-dose: 24 hours/ Multiple-doses: 8 days
  To mearsure the study drug concentration in blood samples which collected after injection
T1/2 of SY-005 following injection of single dose | Single-dose: 24 hours/ Multiple-doses: 8 days
  To mearsure the study drug concentration in blood samples which collected after injection

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided